CLINICAL TRIAL: NCT06647901
Title: Efficacy of ICG-based NIR Imaging in Intralesional Curettage of Giant Cell Tumors of Bone in Limbs: a Prospective, Single-center, Single-arm, Open Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tang Xiaodong (Other)
Responsible Party: Sponsor-Investigator, Tang Xiaodong, Dr., Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-ICGGCT-1
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-05

CONDITIONS: Giant Cell Tumor of Bone
Keywords: ICG; Giant cell tumor of bone; curettage
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICG group (Experimental)
  Interventions: Drug: ICG (Indocyanine Green)

INTERVENTIONS:
Drug: ICG (Indocyanine Green) — Patients will be receive intravenously administrated at a dose of 2 mg/kg on the day before surgery. The drug was dissolved into 250 mL of normal saline and administered using a light-proof infusion apparatus. The time course of administration was 60 min. NIR imaging will be performed during surgery to help identify small tumor residuals.

SUMMARY:
ICG fluorescence imaging will be applied during the intralesional curettage of giant cell tumor of bone in the limbs. This study aims to preliminarily explore whether ICG fluorescent-guided curettage could find small residual tumors and reduce the recurrence rate of tumor.

DETAILED DESCRIPTION:
Recurrence is a problem in the treatment of giant cell tumor of bone(GCTB). With the application of high-speed burr and other adjuvant therapy (phenol, liquid nitrogen freezing, cauterization, etc.), the recurrence rate is greatly reduced, but it is still as high as 20%. The main cause of local recurrence is the difficulty in distinguishing small residual tumor lesions by the naked eye. The application of frozen section is limited due to the long-term decalcification of bone specimens.

Intraoperative near-infrared (NIR) imaging is a promising technology expected to solve the above problems. It allows for real-time scanning of a wide area with tumor showing fluorescence. Such intraoperative fluorescent signals provide objective evidence for the surgeon and are more reliable than subjective visual and tactile information.

This study aims to explore whether ICG-based NIR imaging guided curettage could find small residual tumors and reduce the recurrence rate of GCT.

ELIGIBILITY:
Inclusion Criteria:

1. . Aged 18-65.
2. Biopsy confirmed giant cell tumor of bone.
3. The lesions located in the limbs.
4. This operation is the initial treatment.
5. Denosumab and diphosphonates are not used before surgery.
6. Planned operation is intralesional curettage and filling bone defects with bone cement.
7. Preoperative bone scan and thin layer (layer thickness ≤3.5mm) chest CT plain scan confirmed that the lesion is a single occurrence without metastasis.
8. Subjects fully understand the benefits and risks of this experiment and are still willing to participate and sign the informed consent.

Exclusion Criteria:

1. . Known allergy to iodine contrast, indocyanine green or bone cement.
2. . Severe hepatic and renal insufficiency.
3. . During pregnancy or lactation.
4. . Have other malignant tumors and are receiving related medical treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
local recurrence rate of tumor | From surgery to 2 years after surgery
  To explore whether based on ICG-based-NIR fluorescence imaging assisted intralesional curettage can reduce the local recurrence rate of giant cell tumor of bone in limbs.

SECONDARY OUTCOMES:
Accuracy of ICG prediction tumor residuals | From surgery to 2 weeks after surgery
  To explore the accuracy of ICG fluorescence in detection of small residual tumor lesions and calculate the sensitivity, specificity, positive predictive value, negative predictive value.
Correlation between fluorescence intensity and pathology findings of tumor residuals | From surgery to 2 weeks after surgery
  To explore the correlation between ICG fluorescence intensity and accuracy of detection of residual tumor lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No